CLINICAL TRIAL: NCT02432235
Title: A Phase 1 Adaptive Dose-Escalation Study to Evaluate the Tolerability, Safety, Pharmacokinetics, and Antitumor Activity of ADCT-301 in Patients With Relapsed or Refractory Hodgkin Lymphoma and Non-Hodgkin Lymphoma
Brief Title: Study of ADCT-301 in Patients With Relapsed or Refractory Hodgkin and Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADCT-301-001; 2015-005272-25 (EudraCT Number); 199948 (Registry Identifier: HRA)
Record Dates: First submitted 2015-02-26; First posted 2015-05-04 (Estimated); Results first posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Hodgkin Lymphoma; Non-Hodgkin Lymphoma
Keywords: Camidanlumab tesirine
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Calmodulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (12):
- 3 μg/kg (Experimental): Participants received an intravenous (IV) infusion of camidanlumab tesirine (3 μg/kg) on Day 1 of each 3-week treatment cycle, for a maximum of 2 cycles.
  Interventions: Drug: Camidanlumab tesirine
- 5 μg/kg (Experimental): Participants received an intravenous (IV) infusion of camidanlumab tesirine (5 μg/kg) on Day 1 of each 3-week treatment cycle, for a maximum of 4 cycles.
  Interventions: Drug: Camidanlumab tesirine
- 8 μg/kg (Experimental): Participants received an intravenous (IV) infusion of camidanlumab tesirine (8 μg/kg) on Day 1 of each 3-week treatment cycle, for a maximum of 3 cycles.
  Interventions: Drug: Camidanlumab tesirine
- 13 μg/kg (Experimental): Participants received an intravenous (IV) infusion of camidanlumab tesirine (13 μg/kg) on Day 1 of each 3-week treatment cycle, for a maximum of 15 cycles.
  Interventions: Drug: Camidanlumab tesirine
- 20 μg/kg (Experimental): Participants received an intravenous (IV) infusion of camidanlumab tesirine (20 μg/kg) on Day 1 of each 3-week treatment cycle, for a maximum of 3 cycles.
  Interventions: Drug: Camidanlumab tesirine
- 30 μg/kg (Experimental): Participants received an intravenous (IV) infusion of camidanlumab tesirine (30 μg/kg) on Day 1 of each 3-week treatment cycle, for a maximum of 10 cycles.
  Interventions: Drug: Camidanlumab tesirine
- 45 μg/kg (Experimental): Participants received an intravenous (IV) infusion of camidanlumab tesirine (45 μg/kg) on Day 1 of each 3-week treatment cycle, for a maximum of 10 cycles.
  Interventions: Drug: Camidanlumab tesirine
- 60 μg/kg (Experimental): Participants received an intravenous (IV) infusion of camidanlumab tesirine (60 μg/kg) on Day 1 of each 3-week treatment cycle, for a maximum of 8 cycles.
  Interventions: Drug: Camidanlumab tesirine
- 80 μg/kg (Experimental): Participants received an intravenous (IV) infusion of camidanlumab tesirine (80 μg/kg) on Day 1 of each 3-week treatment cycle, for a maximum of 7 cycles.
  Interventions: Drug: Camidanlumab tesirine
- 100 μg/kg (Experimental): Participants received an intravenous (IV) infusion of camidanlumab tesirine (100 μg/kg) on Day 1 of each 3-week treatment cycle, for a maximum of 5 cycles.
  Interventions: Drug: Camidanlumab tesirine
- 150 μg/kg (Experimental): Participants received an intravenous (IV) infusion of camidanlumab tesirine (150 μg/kg) on Day 1 of each 3-week treatment cycle, for a maximum of 2 cycles.
  Interventions: Drug: Camidanlumab tesirine
- 300 μg/kg (Experimental): A single participant received by error an intravenous (IV) infusion of camidanlumab tesirine (300 μg/kg) on Day 1 of Cycle 1 (planned dose was 30 μg/kg). Dosing in the subsequent cycles was 30 μg/kg (for 2 more cycles).
  Interventions: Drug: Camidanlumab tesirine

INTERVENTIONS:
Drug: Camidanlumab tesirine — Intravenous (IV) infusion.
  Other Names: ADCT-301; Cami

SUMMARY:
This study evaluates camidanlumab tesirine in participants with relapsed/refractory Non-Hodgkin or Hodgkin lymphoma.

DETAILED DESCRIPTION:
This is a Phase I, first in human clinical study with camidanlumab tesirine to evaluate the safety and tolerability and pharmacokinetics of camidanlumab tesirine in participants with relapsed/refractory lymphoma.

Camidanlumab tesirine is a human monoclonal antibody attached via a cleavable linker to a pyrrolobenzodiazepine (PBD) warhead which, when internalized by antigen expressing cells, covalently cross links deoxyribonucleic acid (DNA) preventing replication.

The study will be conducted in 2 parts: Part 1 (dose escalation) and Part 2 (expansion).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 18 years or older.
2. Refractory or relapsed lymphoma (per World Health Organization (WHO) Classification system)
3. Pathologically confirmed relapsed or refractory lymphoma
4. Availability of formalin-fixed paraffin-embedded (FFPE) tumor tissue block.
5. Measurable disease, defined by the 2014 Lugano Classification Criteria and Global Response Score Grading Scales for cutaneous T-cell lymphoma (CTCL)
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
7. Absolute neutrophil count ≥1500/µL. Criterion not applicable to adult T cell leukemia/lymphoma (ATLL) patients.
8. Platelet count of ≥75000/µL. Criterion not applicable to ATLL patients.
9. Hemoglobin ≥9.0 g/dL without transfusion within the 2 weeks prior to Day 1.
10. Serum/plasma creatinine ≤1.5 mg/dL, or if the participant has a creatinine > 1.5 mg/dL, a measured creatinine clearance must be > 80 mL/min as calculated by the Cockcroft and Gault equation
11. Serum alkaline phosphatase, alanine aminotransferase, and aspartate aminotransferase ≤2 times the upper limit of normal (ULN); ≤ 5 times ULN if there is liver or bone involvement.
12. Total serum/plasma bilirubin ≤1.5 times ULN (participants with known Gilbert's syndrome may have a total bilirubin up to ≤3 times ULN)
13. Women of childbearing potential must have a negative serum beta-human chorionic gonadotropin pregnancy test within 7 days prior to Day 1.
14. Women of childbearing potential must agree to use a highly effective method of contraception. Men with female partners who are of childbearing potential must agree that they or their partners will use a highly effective method of contraception.

Exclusion Criteria:

1. Participants who have an option for any treatment with proven clinical benefit for their lymphoid malignancy at current state of disease.
2. Active graft-versus-host disease.
3. Autologous or allogenic transplant within the 60 days prior to Cycle 1 Day 1 (C1D1)
4. Evidence of myelodysplasia or myeloid leukemia by morphology, immunostains, flow cytometry, or cytogenetics on a bone marrow aspirate or biopsy.
5. Known history of positive serum human anti-drug antibody (ADA) or known allergy to any component of ADCT-301.
6. History of symptomatic autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, Sjögren's syndrome, autoimmune vasculitis [e.g., Wegener's granulomatosis])
7. History of neuropathy considered of autoimmune origin (e.g., polyradiculopathy including Guillain-Barré syndrome and myasthenia gravis); other central nervous system autoimmune disease (e.g., poliomyelitis, multiple sclerosis).
8. History of recent infection (within 4 weeks of C1D1) considered to be caused by one of the pathogens listed: herpes simplex virus Type 1 (HSV1), herpes simplex virus Type 2 (HSV2), varicella zoster virus (VZV), Epstein-Barr virus (EBV), cytomegalovirus (CMV), measles, Influenza A, Zika virus, Chikungunya virus, mycoplasma pneumonia, Campylobacter jejuni, or enterovirus D68.
9. Known seropositive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or antibody to hepatitis C virus (anti-HCV) with confirmatory testing and requiring anti-viral therapy. Note: testing is not mandatory to be eligible.

   If participant is at risk for having undiagnosed hepatitis C virus (HCV) (e.g., history of injection drug use), HCV testing should be considered.
10. History of Steven's Johnson's syndrome or toxic epidermal necrolysis syndrome.
11. Pregnant or breastfeeding women.
12. Significant medical comorbidities, including uncontrolled hypertension (diastolic blood pressure > 115 mm Hg), unstable angina, congestive heart failure (greater than New York Heart Association class II), severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia, poorly controlled diabetes, severe chronic pulmonary disease, coronary angioplasty, or myocardial infarction within 6 months prior to screening, or uncontrolled atrial or ventricular cardiac arrhythmias.
13. Use of any other experimental medication(s) within 14 days or 5 half-lives, but in no case < 14 days prior to the start of study treatment on Cycle 1, Day 1, except if approved by the Sponsor.
14. Major surgery, radiotherapy, chemotherapy, or other anti-neoplastic therapy (including prednisone ≥ 40 mg/day or equivalent) within 14 days or 5 half-lives (whichever is shorter) prior to Cycle 1, Day 1 treatment, except if approved by the Sponsor.
15. Failure to recover (to Common Terminology Criteria for Adverse Events [CTCAE Version 4.0] Grade 0 or Grade 1) from acute non-hematologic toxicity (except all grades of alopecia or Grade 2 or lower neuropathy), due to previous therapy, prior to Screening.
16. Congenital long QT syndrome or a corrected QT interval (QTc)≥ 450 ms at screening (unless secondary to pacemaker or bundle branch block).
17. Active second primary malignancy other than non-melanoma skin cancers, nonmetastatic prostate cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast, or other malignancy that Sponsor Medical Monitor and Investigator agree, and document should not be exclusionary.
18. Any other significant medical illness, abnormality, or condition that would, in the Investigator's judgment, make the participant inappropriate for study participation or put the participant at risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2019-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Wuerthner, MD, PhD, Study Director — ADC Therapeutics
Locations (12):
- United States (7):
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The University of Texas/MD Anderson Cancer Center, Houston, Texas
  - Cancer Therapy and Research Center at The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Froedtert Hospital/Medical College of Wisconsin, Milwaukee, Wisconsin
- United Kingdom (5):
  - Guy's and St. Thomas' Hospital NHS Trust, London, England
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, England
  - Churchill Hospital, Oxford University Hospitals NHS Foundation Trust, Oxford, England
  - The Christie NHS Foundation Trust, Manchester, Greater Manchester
  - Southampton General Hospital, University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toukam M, Wuerthner J, Havenith K, Hamadani M, Caimi PF, Kopotsha T, Cruz HG, Boni JP. Population pharmacokinetics analysis of camidanlumab tesirine in patients with relapsed or refractory Hodgkin lymphoma and non-Hodgkin lymphoma. Cancer Chemother Pharmacol. 2023 Jan;91(1):13-24. doi: 10.1007/s00280-022-04486-4. Epub 2022 Nov 4. PMID 36333464
- [Derived] Toukam M, Boni JP, Hamadani M, Caimi PF, Cruz HG, Wuerthner J. Exposure-response analysis of Camidanlumab tesirine in patients with relapsed or refractory classical Hodgkin lymphoma and non-Hodgkin lymphoma. Cancer Chemother Pharmacol. 2023 Jan;91(1):1-12. doi: 10.1007/s00280-022-04487-3. Epub 2022 Nov 4. PMID 36333463
- [Derived] Hamadani M, Collins GP, Caimi PF, Samaniego F, Spira A, Davies A, Radford J, Menne T, Karnad A, Zain JM, Fields P, Havenith K, Cruz HG, He S, Boni J, Feingold J, Wuerthner J, Horwitz S. Camidanlumab tesirine in patients with relapsed or refractory lymphoma: a phase 1, open-label, multicentre, dose-escalation, dose-expansion study. Lancet Haematol. 2021 Jun;8(6):e433-e445. doi: 10.1016/S2352-3026(21)00103-4. PMID 34048682

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 12 sites that screened and enrolled participants: USA: 7 sites; UK: 5 sites.
Pre-assignment Details: Participants were included in a screening period of up to 28 days.
Period: Overall Study
Arm/Group | 3 μg/kg | 5 μg/kg | 8 μg/kg | 13 μg/kg | 20 μg/kg | 30 μg/kg | 45 μg/kg | 60 μg/kg | 80 μg/kg | 100 μg/kg | 150 μg/kg | 300 μg/kg
Started | 2 | 2 | 2 | 3 | 2 | 20 | 41 | 29 | 26 | 3 | 2 | 1
Completed | 1 | 0 | 0 | 1 | 0 | 8 | 23 | 9 | 5 | 0 | 1 | 0
Not Completed | 1 | 2 | 2 | 2 | 2 | 12 | 18 | 20 | 21 | 3 | 1 | 1
Not completed — Death | 1 | 1 | 2 | 2 | 1 | 3 | 11 | 15 | 15 | 3 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 2 | 5 | 3 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Miscellaneous | 0 | 0 | 0 | 0 | 1 | 6 | 2 | 2 | 4 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3 μg/kg | 5 μg/kg | 8 μg/kg | 13 μg/kg | 20 μg/kg | 30 μg/kg | 45 μg/kg | 60 μg/kg | 80 μg/kg | 100 μg/kg | 150 μg/kg | 300 μg/kg | Total
Number analyzed (Participants) | 2 | 2 | 2 | 3 | 2 | 20 | 41 | 29 | 26 | 3 | 2 | 1 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.5 (2.12) | 44.0 (2.83) | 64.0 (12.73) | 51.0 (12.53) | 38.0 (19.80) | 42.1 (16.32) | 45.1 (15.48) | 56.3 (18.16) | 58.1 (15.69) | 58.7 (8.08) | 44.5 (19.09) | 64.0 | 50.8 (17.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 2 | 1 | 8 | 14 | 15 | 10 | 0 | 1 | 1 | 55
  Male | 1 | 1 | 1 | 1 | 1 | 12 | 27 | 14 | 16 | 3 | 1 | 0 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 2 | 5 | 3 | 2 | 0 | 0 | 0 | 13
  Not Hispanic or Latino | 2 | 1 | 2 | 3 | 2 | 18 | 36 | 26 | 24 | 3 | 2 | 1 | 120
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 0 | 0 | 5 | 1 | 9 | 0 | 0 | 0 | 17
  White | 1 | 2 | 2 | 1 | 1 | 19 | 30 | 28 | 17 | 2 | 2 | 1 | 106
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 2 | 3 | 2 | 20 | 27 | 20 | 16 | 2 | 1 | 1 | 98
  United Kingdom | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 9 | 10 | 1 | 1 | 0 | 35
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status was graded on a scale of 0-5, where a higher score indicated a worse outcome:
  0. = fully active
  1. = capable of light work of a sedentary nature
  2. = capable of self-care; unable to carry out work activities
  3. = capable of only limited self-care
  4. = completely disabled; cannot carry out any self-care
  5. = dead
  Participants
    Grade 0 | 0 | 1 | 0 | 0 | 0 | 6 | 16 | 12 | 7 | 0 | 1 | 0 | 43
    Grade 1 | 2 | 0 | 2 | 1 | 2 | 14 | 24 | 13 | 16 | 3 | 1 | 1 | 79
    Grade 2 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 4 | 3 | 0 | 0 | 0 | 11
    Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 98.05 (26.517) | 55.25 (12.799) | 80.40 (19.658) | 63.57 (4.840) | 65.05 (14.496) | 79.18 (19.920) | 89.10 (31.926) | 75.15 (18.241) | 78.19 (15.780) | 82.67 (15.808) | 96.50 (12.869) | 53.20 | 80.69 (23.766)
Height [Mean (Standard Deviation); unit: centimeters (cm)] — Population: One participant in the 20 μg/kg group, one participant in the 30 μg/kg group and two participants in the 45 μg/kg group did not have their height measurement taken.
  centimeters (cm)
    number analyzed (Participants) | 2 | 2 | 2 | 3 | 1 | 19 | 39 | 29 | 26 | 3 | 2 | 1 | 129
    (all) | 176.65 (24.961) | 158.00 (1.414) | 176.00 (4.243) | 170.43 (5.811) | 170.20 | 172.13 (11.212) | 172.12 (9.410) | 171.43 (9.341) | 170.33 (10.188) | 173.43 (10.856) | 172.50 (13.435) | 155.00 | 171.37 (9.920)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: One participant in the 20 μg/kg group, one participant in the 30 μg/kg group and two participants in the 45 μg/kg group did not have their height measurement taken, and so their Body Mass Index could not be calculated.
  kg/m^2
    number analyzed (Participants) | 2 | 2 | 2 | 3 | 1 | 19 | 39 | 29 | 26 | 3 | 2 | 1 | 129
    (all) | 33.60 (17.816) | 22.18 (5.524) | 25.83 (5.100) | 21.98 (2.829) | 25.99 | 26.69 (4.496) | 30.26 (11.193) | 25.37 (4.913) | 26.95 (4.944) | 27.47 (4.559) | 33.07 (9.447) | 22.14 | 27.52 (7.757)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: A DLT defined as any of the following, except those that are clearly due to underlying disease or extraneous causes:
  A hematologic DLT is defined as (different considerations for Adult T-Cell Leukemia/Lymphoma (ATLL) participants):
  * Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 or 4 febrile neutropenia or neutropenic infection
  * CTCAE Grade 4 neutropenia lasting >7 days
  * CTCAE Grade 4 thrombocytopenia
  * CTCAE Grade 3 thrombocytopenia with clinically significant bleeding, or Grade 3 thrombocytopenia requiring a platelet transfusion
  * CTCAE Grade 4 anemia
  A non-hematologic DLT is defined as:
  * CTCAE Grade 4 tumor lysis syndrome
  * CTCAE Grade 3 or higher AE (including nausea, vomiting, diarrhea, electrolyte imbalances lasting ≥ 48 hours despite optimal therapy; excluding all grades of alopecia)
  * CTCAE Grade 3 or higher hypersensitivity reaction
  * CTCAE Grade 2 or higher skin ulceration
  * CTCAE Grade 2 or higher peripheral sensory or motor neuropathy
Time Frame: Cycle 1 Day 1 to end of Cycle 1 or 2 (21 day cycle length)
Population: DLT Evaluable Analysis Set: The DLT-evaluable analysis set consisted of participants who completed two cycles of ADCT-301 if enrolled prior to protocol amendment 4 and participants who completed one cycle of ADCT-301 if enrolled after protocol amendment 4. The participants with completed DLT information were included even if they discontinued early before the end of cycle 2 or cycle 1 respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | 3 μg/kg | 5 μg/kg | 8 μg/kg | 13 μg/kg | 20 μg/kg | 30 μg/kg | 45 μg/kg | 60 μg/kg | 80 μg/kg | 100 μg/kg | 150 μg/kg | 300 μg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 10 | 15 | 29 | 16 | 3 | 2 | 1
Participants | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0

2. Primary Outcome: Recommended Dose of Camidanlumab Tesirine for Part 2
Description: The recommended dose was established by the dose escalation steering committee and based on safety findings during Part 1 of the study.
Time Frame: Cycle 1 Day 1 to end of Cycle 1 or 2 (21 day cycle length)
Population: Number of participants analyzed presented in the outcome measure data are only those participants in the DLT evaluable analysis set who were dosed at the three dose levels recommended for Part 2.
Measure: Number; unit: μg/kg
Groups:
- Dose-Limiting Toxicity (DLT) Evaluable Set Analysis Set: DLT Evaluable Analysis Set: The DLT-evaluable analysis set consisted of participants who completed two cycles of ADCT-301 if enrolled prior to protocol amendment 4 and participants who completed one cycle of ADCT-301 if enrolled after protocol amendment 4. The participants with completed DLT information were included even if they discontinued early before the end of cycle 2 or cycle 1 respectively.
Arm/Group | Dose-Limiting Toxicity (DLT) Evaluable Set Analysis Set
Number analyzed (Participants) | 86
μg/kg
  Participants with Hodgkin Lymphoma (Dose level 1: 30 µg/kg): number analyzed (Participants) | 10
  Participants with Hodgkin Lymphoma (Dose level 1: 30 µg/kg) | 30
  Participants with Hodgkin Lymphoma (Dose level 2: 45 µg/kg): number analyzed (Participants) | 15
  Participants with Hodgkin Lymphoma (Dose level 2: 45 µg/kg) | 45
  Participants with T-cell Lymphoma (80 µg/kg): number analyzed (Participants) | 16
  Participants with T-cell Lymphoma (80 µg/kg) | 80

3. Primary Outcome: Number of Participants Reporting at Least One Treatment Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant enrolled into this study regardless of its causal relationship to study drug. A TEAE is defined as any event not present before exposure to study drug or any event already present that worsens in either intensity or frequency after exposure to study drug.
Time Frame: Day 1 up to 84 days after last dose (median time on treatment was 43 days [min 1 day; max 354 days])
Measure: Count of Participants; unit: Participants
Arm/Group | 3 μg/kg | 5 μg/kg | 8 μg/kg | 13 μg/kg | 20 μg/kg | 30 μg/kg | 45 μg/kg | 60 μg/kg | 80 μg/kg | 100 μg/kg | 150 μg/kg | 300 μg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 3 | 2 | 20 | 41 | 29 | 26 | 3 | 2 | 1
Participants | 1 | 2 | 2 | 3 | 2 | 20 | 41 | 29 | 26 | 3 | 2 | 1

4. Primary Outcome: Number of Participants Reporting at Least One Treatment Emergent Serious Adverse Event (SAE)
Description: A treatment-emergent AE (TEAE) is defined as any event not present before exposure to study drug or any event already present that worsens in either intensity or frequency after exposure to study drug. An SAE is defined as any event that results in death, is immediately life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.
Time Frame: Day 1 up to 84 days after last dose (median time on treatment was 43 days [min 1 day; max 354 days])
Measure: Count of Participants; unit: Participants
Arm/Group | 3 μg/kg | 5 μg/kg | 8 μg/kg | 13 μg/kg | 20 μg/kg | 30 μg/kg | 45 μg/kg | 60 μg/kg | 80 μg/kg | 100 μg/kg | 150 μg/kg | 300 μg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 3 | 2 | 20 | 41 | 29 | 26 | 3 | 2 | 1
Participants | 0 | 1 | 0 | 3 | 1 | 10 | 24 | 14 | 18 | 1 | 1 | 1

5. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the number of participants with a best overall response of complete response (CR) or partial response (PR) at the time each participant discontinued treatment with camidanlumab tesirine.
  Tumor response was assessed using the 2014 Lugano Classification.
  CR is defined as achieving each of the following:
  * Complete metabolic response.
  * Complete radiologic response (target node regress to <1.5 cm, no nonmeasured lesions, no organ enlargement, no new lesions and normal bone marrow morphology).
  PR is defined as achieving each of the following:
  * Partial metabolic response (findings indicate residual disease).
  * Partial remission (>50% decrease in target measurable nodes, regression/ absence/ no increase of nonmeasured lesions, spleen regressed by >50% in length and no new lesions).
Time Frame: Day 1 to End of Study (a maximum of 12 months after treatment; median time on treatment was 43 days [min 1 day; max 354 days])
Population: Efficacy Analysis Set: The efficacy analysis set consisted of participants who received at least one dose of camidanlumab tesirine with a valid baseline and at least one valid post-baseline disease assessment or participants who had documented progression of disease or death at any time after the first dose of study.
Measure: Count of Participants; unit: Participants
Arm/Group | 3 μg/kg | 5 μg/kg | 8 μg/kg | 13 μg/kg | 20 μg/kg | 30 μg/kg | 45 μg/kg | 60 μg/kg | 80 μg/kg | 100 μg/kg | 150 μg/kg | 300 μg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 3 | 2 | 20 | 41 | 28 | 24 | 3 | 2 | 1
Participants | 0 | 0 | 0 | 1 | 0 | 11 | 32 | 15 | 12 | 2 | 1 | 1

6. Secondary Outcome: Duration of Response (DoR)
Description: DoR is defined among responders (complete response [CR] and partial response [PR]) as the time from the earliest date of first response until the first date of either disease progression or death due to any cause. Tumor response was assessed using the 2014 Lugano Classification.
  Disease progression is defined as progressive metabolic disease and one of the follow:
  * Target node progression.
  * An individual extranodal lesion must be abnormal with length > 1.5cm and/or increase of length > 50%.
  * New or clear progression of nonmeasured lesions.
  * Regrowth of previously resolved lesions or new nodes >1.5 cm in length.
  * New or recurrent bone marrow involvement.
  DoR is presented overall for all participants who were classed as responders among the efficacy analysis set. Data is pooled for all lymphoma participants for DoR as specified in protocol section 8.4.
Time Frame: Day 1 to End of Study (a maximum of 12 months after last dose; median time on treatment was 43 days [min 1 day; max 354 days])
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Efficacy Analysis Set: Participants received an intravenous (IV) infusion of camidanlumab tesirine at any dose (doses ranging from 3 μg/kg to 300 μg/kg) on Day 1 of each 3-week treatment cycle. The maximum number of cycles received was 15.
Arm/Group | Efficacy Analysis Set
Number analyzed (Participants) | 130
Months | 5.19 [4.50 to 7.23]

7. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival (PFS) is defined among the efficacy population as the time from first dose of study drug until either disease progression or death due to any cause. Tumor response was assessed using the 2014 Lugano Classification for response.
  Disease progression is defined as progressive metabolic disease and one of the following:
  * Target node progression.
  * An individual extranodal lesion must be abnormal with length > 1.5cm and/or increase of length > 50%.
  * New or clear progression of nonmeasured lesions.
  * Regrowth of previously resolved lesions or new nodes > 1.5 cm in length.
  * New or recurrent bone marrow involvement.
  PFS is presented overall for all participants who received camidanlumab tesirine among the efficacy analysis set. Data is pooled for all lymphoma participants for PFS as specified in protocol section 8.4
Time Frame: as for outcome 6
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Efficacy Analysis Set
Number analyzed (Participants) | 130
Months | 5.22 [3.78 to 5.95]

8. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from the first dose of study drug treatment until the date of death due to any cause.
  OS is presented overall for all participants who received camidanlumab tesirine among the efficacy analysis set. Data is pooled for all lymphoma participants for OS as specified in protocol section 8.4.
Time Frame: as for outcome 6
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Efficacy Analysis Set
Number analyzed (Participants) | 130
Months | 16.26 [10.02 to NA] — Insufficient number of participants died during the study, so confidence upper limit could not be calculated.

9. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) for Camidanlumab Tesirine
Description: Cmax for HuMax-TAC, pyrrolobenzodiazepine (PBD) conjugated HuMax-TAC, and free warhead (SG3199).
Time Frame: Pre-dose on Day 1 and 1 to 336 hours post-dose of Cycles 1 and 2 (21 day cycle length)
Population: Pharmacokinetic (PK) analysis set consisted of all participants who received study drug and have sufficient concentration data for PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 3 μg/kg | 5 μg/kg | 8 μg/kg | 13 μg/kg | 20 μg/kg | 30 μg/kg | 45 μg/kg | 60 μg/kg | 80 μg/kg | 100 μg/kg | 150 μg/kg | 300 μg/kg
Number analyzed (Participants) | 1 | 1 | 2 | 3 | 2 | 20 | 41 | 29 | 25 | 3 | 2 | 1
ng/mL
  Cycle 1 - HuMax-TAC: number analyzed (Participants) | 1 | 1 | 2 | 3 | 2 | 20 | 41 | 28 | 23 | 3 | 2 | 1
  Cycle 1 - HuMax-TAC | 109 | 62.5 | 131 (20.7) | 189 (98.4) | 318 (82.9) | 603 (31.8) | 803 (54.4) | 1120 (82.8) | 1325 (43.1) | 1494 (26.1) | 2671 (32.9) | 5020
  Cycle 2 - HuMax-TAC: number analyzed (Participants) | 1 | 0 | 2 | 2 | 1 | 19 | 35 | 23 | 16 | 2 | 2 | 1
  Cycle 2 - HuMax-TAC | 67.5 |  | 177 (39.4) | 254 (13.1) | 224 | 554 (48.1) | 1040 (60.0) | 1402 (56.1) | 1379 (32.2) | 800 (726) | 3251 (37.8) | 497
  Cycle 1 - PBD-conjugated HuMax-TAC: number analyzed (Participants) | 1 | 0 | 2 | 3 | 2 | 20 | 41 | 29 | 25 | 3 | 2 | 1
  Cycle 1 - PBD-conjugated HuMax-TAC | 79.5 |  | 127 (27.6) | 152 (95.1) | 241 (76.7) | 455 (38.5) | 648 (51.0) | 881 (78.8) | 1055 (45.9) | 1154 (26.4) | 2097 (21.1) | 4020
  Cycle 2 - PBD-conjugated HuMax-TAC: number analyzed (Participants) | 1 | 0 | 2 | 2 | 1 | 19 | 35 | 23 | 17 | 2 | 2 | 1
  Cycle 2 - PBD-conjugated HuMax-TAC | 61.5 |  | 151 (23.2) | 208 (18.4) | 164 | 424 (47.8) | 808 (55.8) | 1084 (59.9) | 1084 (32.0) | 645 (655) | 2090 (31.6) | 497
  Cycle 1 - Free warhead (SG3199): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 4 | 12 | 1 | 1 | 1
  Cycle 1 - Free warhead (SG3199) |  |  |  |  |  |  | 0.0120 (8.04) | 0.0310 (102) | 0.0150 (34.6) | 0.0110 | 0.0170 | 0.0240
  Cycle 2 - Free warhead (SG3199): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 3 | 1 | 2 | 0
  Cycle 2 - Free warhead (SG3199) |  |  |  |  |  |  | 0.0170 (46.9) | 0.132 (413) | 0.0140 (4.21) | 0.0270 | 0.0170 (20.1) |

10. Secondary Outcome: Time to Reach the Maximum Serum Concentration (Tmax) for Camidanlumab Tesirine
Description: Tmax for HuMax-TAC, PBD-conjugated HuMax-TAC, and free warhead (SG3199).
Time Frame: Pre-dose on Day 1 and 1 to 336 hours post-dose of Cycles 1 and 2 (21 day cycle length)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | 3 μg/kg | 5 μg/kg | 8 μg/kg | 13 μg/kg | 20 μg/kg | 30 μg/kg | 45 μg/kg | 60 μg/kg | 80 μg/kg | 100 μg/kg | 150 μg/kg | 300 μg/kg
Number analyzed (Participants) | 1 | 1 | 2 | 3 | 2 | 20 | 41 | 29 | 25 | 3 | 2 | 1
Days
  Cycle 1 - HuMax-TAC: number analyzed (Participants) | 1 | 1 | 2 | 3 | 2 | 20 | 41 | 28 | 23 | 3 | 2 | 1
  Cycle 1 - HuMax-TAC | 0.155 | 0.0830 | 0.0970 (22.4) | 0.149 (75.3) | 0.103 (26.4) | 0.0820 (38.5) | 0.0950 (67.5) | 0.106 (58.3) | 0.105 (45.1) | 0.111 (22.3) | 0.157 (0.937) | 0.172
  Cycle 2 - HuMax-TAC: number analyzed (Participants) | 1 | 0 | 2 | 2 | 1 | 19 | 35 | 23 | 16 | 2 | 2 | 1
  Cycle 2 - HuMax-TAC | 0.149 |  | 0.110 (32.2) | 0.137 (69.8) | 0.130 | 0.0640 (105) | 0.0790 (81.6) | 0.0910 (100) | 0.0830 (71.7) | 0.0700 (31.4) | 0.145 (21.1) | 0.0310
  Cycle 1 - PBD-conjugated HuMax-TAC: number analyzed (Participants) | 1 | 0 | 2 | 3 | 2 | 20 | 41 | 29 | 25 | 3 | 2 | 1
  Cycle 1 - PBD-conjugated HuMax-TAC | 0.155 |  | 0.114 (46.4) | 0.110 (24.6) | 0.131 (64.3) | 0.0910 (47.1) | 0.0950 (62.4) | 0.0970 (44.6) | 0.118 (83.0) | 0.111 (22.3) | 0.114 (46.7) | 0.0830
  Cycle 2 - PBD-conjugated HuMax-TAC: number analyzed (Participants) | 1 | 0 | 2 | 2 | 1 | 19 | 35 | 23 | 17 | 2 | 2 | 1
  Cycle 2 - PBD-conjugated HuMax-TAC | 0.336 |  | 0.126 (37.9) | 0.0860 (1.70) | 0.0920 | 0.0640 (121) | 0.0660 (64.3) | 0.0690 (110) | 0.0720 (79.3) | 0.0850 (2.89) | 0.0940 (160) | 0.0310
  Cycle 1 - Free warhead (SG3199): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 4 | 12 | 1 | 1 | 1
  Cycle 1 - Free warhead (SG3199) |  |  |  |  |  |  | 0.119 (75.0) | 0.124 (83.6) | 0.206 (69.8) | 0.211 | 0.240 | 0.172
  Cycle 2 - Free warhead (SG3199): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 3 | 1 | 2 | 0
  Cycle 2 - Free warhead (SG3199) |  |  |  |  |  |  | 0.192 (42.6) | 0.0970 (119) | 0.201 (24.8) | 0.167 | 0.156 (109) |

11. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-last) for Camidanlumab Tesirine
Description: AUC0-last for HuMax-TAC, PBD-conjugated HuMax-TAC, and free warhead (SG3199).
Time Frame: Pre-dose on Day 1 and 1 to 336 hours post-dose of Cycles 1 and 2 (21 day cycle length)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | 3 μg/kg | 5 μg/kg | 8 μg/kg | 13 μg/kg | 20 μg/kg | 30 μg/kg | 45 μg/kg | 60 μg/kg | 80 μg/kg | 100 μg/kg | 150 μg/kg | 300 μg/kg
Number analyzed (Participants) | 1 | 1 | 2 | 3 | 2 | 20 | 41 | 29 | 25 | 3 | 2 | 1
day*ng/mL
  Cycle 1 - HuMax-TAC: number analyzed (Participants) | 1 | 1 | 2 | 3 | 2 | 20 | 41 | 28 | 23 | 3 | 2 | 1
  Cycle 1 - HuMax-TAC | 82.7 | 2.60 | 48.2 (207) | 76.3 (1444) | 660 (93.7) | 967 (60.4) | 1715 (128) | 2491 (132) | 2751 (109) | 4091 (84.6) | 12919 (14.6) | 30759
  Cycle 2 - HuMax-TAC: number analyzed (Participants) | 1 | 0 | 2 | 3 | 1 | 19 | 35 | 23 | 16 | 2 | 2 | 1
  Cycle 2 - HuMax-TAC | 21.0 |  | 111 (35.0) | 453 (35.3) | 473 | 1004 (66.8) | 2476 (117) | 3665 (127) | 4190 (123) | 921 (1700356) | 12767 (13.1) | 919
  Cycle 1 - PBD-conjugated HuMax-TAC: number analyzed (Participants) | 1 | 0 | 2 | 3 | 2 | 20 | 41 | 29 | 25 | 3 | 2 | 1
  Cycle 1 - PBD-conjugated HuMax-TAC | 12.0 |  | 58.8 (458) | 76.8 (470) | 262 (276) | 625 (53.1) | 1173 (113) | 1623 (102) | 1630 (155) | 2849 (68.0) | 7727 (11.2) | 18915
  Cycle 2 - PBD-conjugated HuMax-TAC: number analyzed (Participants) | 1 | 0 | 2 | 2 | 1 | 19 | 35 | 23 | 17 | 2 | 2 | 1
  Cycle 2 - PBD-conjugated HuMax-TAC | 18.6 |  | 85.8 (15.9) | 237 (23.1) | 330 | 655 (53.3) | 1514 (103) | 2283 (94.5) | 3038 (97.7) | 1482 (13082) | 8992 (28.3) | 634
  Cycle 1 - Free warhead (SG3199): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 4 | 12 | 1 | 1 | 1
  Cycle 1 - Free warhead (SG3199) |  |  |  |  |  |  | 0.00200 (331) | 0.00200 (127) | 0.00300 (290) | 0.0100 | 0.00400 | 0.0360
  Cycle 2 - Free warhead (SG3199): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 3 | 1 | 2 | 0
  Cycle 2 - Free warhead (SG3199) |  |  |  |  |  |  | 0.00300 (74.6) | 0.0330 (183) | 0.00600 (79.8) | 0.00300 | 0.0130 (5.60) |

12. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time 0 to the End of the Dosing Interval (AUC0-t) for Camidanlumab Tesirine
Description: AUC0-tau for HuMax-TAC, PBD-conjugated HuMax-TAC, and free warhead (SG3199) for Cycle 2 only.
Time Frame: Pre-dose on Day 1 and 1 to 336 hours post-dose of Cycle 2 (21 day cycle length)
Population: as for outcome 9
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | 3 μg/kg | 5 μg/kg | 8 μg/kg | 13 μg/kg | 20 μg/kg | 30 μg/kg | 45 μg/kg | 60 μg/kg | 80 μg/kg | 100 μg/kg | 150 μg/kg | 300 μg/kg
Number analyzed (Participants) | 0 | 0 | 2 | 2 | 1 | 18 | 33 | 23 | 17 | 2 | 2 | 1
day*ng/mL
  Cycle 2 - HuMax-TAC: number analyzed (Participants) | 0 | 0 | 2 | 2 | 1 | 18 | 33 | 23 | 17 | 1 | 2 | 1
  Cycle 2 - HuMax-TAC |  |  | 195 (22.3) | 596 (25.9) | 747 | 1384 (62.6) | 3604 (68.9) | 4688 (98.3) | 5689 (58.2) | 18830 | 17031 (45.1) | 1074
  Cycle 2 - PBD-conjugated HuMax-TAC: number analyzed (Participants) | 0 | 0 | 1 | 2 | 1 | 18 | 33 | 23 | 17 | 2 | 2 | 1
  Cycle 2 - PBD-conjugated HuMax-TAC |  |  | 185 | 385 (28.5) | 489 | 939 (53.6) | 2183 (61.6) | 2811 (76.7) | 3469 (91.3) | 1809 (4154) | 9851 (28.3) | 763
  Cycle 2 - Free warhead (SG3199): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Cycle 2 - Free warhead (SG3199) |  |  |  |  |  |  |  |  |  |  | 0.0310 |

13. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time 0 to Infinity (AUC∞) for Camidanlumab Tesirine
Description: AUC∞ HuMax-TAC and PBD-conjugated HuMax-TAC for Cycle 1 only.
Time Frame: Pre-dose on Day 1 and 1 to 336 hours post-dose of Cycle 1 (21 day cycle length)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | 3 μg/kg | 5 μg/kg | 8 μg/kg | 13 μg/kg | 20 μg/kg | 30 μg/kg | 45 μg/kg | 60 μg/kg | 80 μg/kg | 100 μg/kg | 150 μg/kg | 300 μg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 14 | 29 | 23 | 18 | 2 | 2 | 1
day*ng/mL
  Cycle 1 - HuMax-TAC: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 23 | 23 | 18 | 2 | 2 | 1
  Cycle 1 - HuMax-TAC |  |  |  |  |  | 1283 (63.1) | 3001 (75.0) | 3618 (52.9) | 3261 (83.9) | 4972 (116) | 13842 (9.45) | 33153
  Cycle 1 - PBD-conjugated HuMax-TAC: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 7 | 29 | 19 | 17 | 2 | 2 | 1
  Cycle 1 - PBD-conjugated HuMax-TAC |  |  |  |  | 917 | 1019 (54.9) | 1846 (59.9) | 2284 (50.8) | 2797 (81.7) | 3734 (82.7) | 8730 (5.31) | 20144

14. Secondary Outcome: Accumulation Index (AI) for Camidanlumab Tesirine
Description: AI for HuMax-TAC, PBD-conjugated HuMax-TAC, and free warhead (SG3199). AI is the ratio of area under the serum concentration-time curve (AUC) from 0 to 21 days for Cycle 2 divided by AUC from 0 to 21 days for Cycle 1 (21 day cycle length). It is the increase in drug plasma concentration after multiple dosing until a steady state is reached.
Time Frame: Pre-dose on Day 1 and 1 to 336 hours post-dose of Cycles 1 and 2 (21 day cycle length)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | 3 μg/kg | 5 μg/kg | 8 μg/kg | 13 μg/kg | 20 μg/kg | 30 μg/kg | 45 μg/kg | 60 μg/kg | 80 μg/kg | 100 μg/kg | 150 μg/kg | 300 μg/kg
Number analyzed (Participants) | 0 | 0 | 2 | 2 | 1 | 18 | 33 | 22 | 17 | 2 | 2 | 1
Ratio
  HuMax-TAC: number analyzed (Participants) | 0 | 0 | 2 | 2 | 1 | 16 | 33 | 21 | 15 | 1 | 2 | 1
  HuMax-TAC |  |  | 1.00 (0.0000132) | 1.00 (0.000584) | 1.00 | 1.01 (3.41) | 1.02 (2.59) | 1.03 (4.24) | 1.04 (3.48) | 1.23 | 1.08 (6.58) | 1.00
  PBD-conjugated HuMax-TAC: number analyzed (Participants) | 0 | 0 | 1 | 2 | 1 | 18 | 30 | 22 | 17 | 2 | 2 | 1
  PBD-conjugated HuMax-TAC |  |  | 1.00 | 1.00 (0.00153) | 1.00 | 1.00 (0.234) | 1.01 (1.48) | 1.03 (4.94) | 1.03 (2.38) | 1.06 (8.36) | 1.06 (0.381) | 1.00
  Free warhead (SG3199): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Free warhead (SG3199) |  |  |  |  |  |  |  |  |  |  | 1.00 |

15. Secondary Outcome: Volume of Distribution for Camidanlumab Tesirine
Description: Volume of distribution for HuMax-TAC, PBD-conjugated HuMax-TAC, and free warhead (SG3199).
Time Frame: Pre-dose on Day 1 and 1 to 336 hours post-dose of Cycles 1 and 2 (21 day cycle length)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | 3 μg/kg | 5 μg/kg | 8 μg/kg | 13 μg/kg | 20 μg/kg | 30 μg/kg | 45 μg/kg | 60 μg/kg | 80 μg/kg | 100 μg/kg | 150 μg/kg | 300 μg/kg
Number analyzed (Participants) | 0 | 0 | 2 | 2 | 1 | 18 | 33 | 23 | 18 | 2 | 2 | 1
Liters
  Cycle 1 - HuMax-TAC: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 23 | 23 | 18 | 2 | 2 | 1
  Cycle 1 - HuMax-TAC |  |  |  |  |  | 3.93 (43.2) | 4.57 (26.9) | 4.55 (27.0) | 4.28 (159) | 6.11 (8.73) | 7.01 (46.4) | 4.84
  Cycle 2 - HuMax-TAC: number analyzed (Participants) | 0 | 0 | 2 | 2 | 1 | 16 | 33 | 21 | 15 | 1 | 2 | 1
  Cycle 2 - HuMax-TAC |  |  | 3.71 (70.3) | 3.26 (19.9) | 7.72 | 4.28 (60.1) | 4.54 (36.0) | 4.64 (26.5) | 5.23 (24.8) | 5.55 | 6.13 (6.58) | 2.44
  Cycle 1 - PBD-conjugated HuMax-TAC: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 7 | 29 | 19 | 17 | 2 | 2 | 1
  Cycle 1 - PBD-conjugated HuMax-TAC |  |  |  |  | 2.23 | 3.28 (56.7) | 5.08 (23.3) | 5.05 (25.5) | 5.15 (34.5) | 6.91 (14.4) | 9.03 (71.7) | 5.84
  Cycle 2 - PBD-conjugated HuMax-TAC: number analyzed (Participants) | 0 | 0 | 1 | 2 | 1 | 18 | 30 | 22 | 17 | 2 | 2 | 1
  Cycle 2 - PBD-conjugated HuMax-TAC |  |  | 5.89 | 3.56 (14.7) | 8.39 | 4.81 (53.0) | 4.91 (29.9) | 5.10 (30.2) | 5.89 (25.7) | 14.5 (257) | 7.55 (8.86) | 2.90
  Cycle 2 - Free warhead (SG3199): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Cycle 2 - Free warhead (SG3199) |  |  |  |  |  |  |  |  |  |  | 7246 |

16. Secondary Outcome: Apparent Terminal Half-life (T1/2) of Camidanlumab Tesirine
Description: T1/2 of HuMax-TAC, PBD-conjugated HuMax-TAC, and free warhead (SG3199).
Time Frame: Pre-dose on Day 1 and 1 to 336 hours post-dose of Cycles 1 and 2 (21 day cycle length)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | 3 μg/kg | 5 μg/kg | 8 μg/kg | 13 μg/kg | 20 μg/kg | 30 μg/kg | 45 μg/kg | 60 μg/kg | 80 μg/kg | 100 μg/kg | 150 μg/kg | 300 μg/kg
Number analyzed (Participants) | 0 | 0 | 2 | 2 | 1 | 18 | 33 | 23 | 18 | 2 | 2 | 1
Days
  Cycle 1 - HuMax-TAC: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 23 | 23 | 18 | 2 | 2 | 1
  Cycle 1 - HuMax-TAC |  |  |  |  |  | 1.58 (58.9) | 2.62 (44.1) | 2.76 (51.9) | 1.98 (78.1) | 2.49 (131) | 4.42 (0.622) | 7.68
  Cycle 2 - HuMax-TAC: number analyzed (Participants) | 0 | 0 | 2 | 2 | 1 | 16 | 33 | 21 | 15 | 1 | 2 | 1
  Cycle 2 - HuMax-TAC |  |  | 0.835 (16.9) | 1.63 (0.507) | 2.61 | 1.87 (50.7) | 3.26 (38.0) | 3.26 (59.5) | 3.65 (42.4) | 8.74 | 5.38 (34.4) | 1.43
  Cycle 1 - PBD-conjugated HuMax-TAC: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 7 | 29 | 19 | 17 | 2 | 2 | 1
  Cycle 1 - PBD-conjugated HuMax-TAC |  |  |  |  | 1.75 | 1.39 (49.8) | 2.31 (45.5) | 2.43 (44.7) | 2.11 (78.6) | 2.92 (152) | 5.59 (50.9) | 7.16
  Cycle 2 - PBD-conjugated HuMax-TAC: number analyzed (Participants) | 0 | 0 | 1 | 2 | 1 | 18 | 30 | 22 | 17 | 2 | 2 | 1
  Cycle 2 - PBD-conjugated HuMax-TAC |  |  | 1.30 | 1.37 (5.69) | 2.24 | 1.78 (28.4) | 2.69 (40.2) | 2.93 (62.2) | 3.06 (67.2) | 3.03 (156) | 5.02 (2.26) | 1.67
  Cycle 2 - Free warhead (SG3199): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Cycle 2 - Free warhead (SG3199) |  |  |  |  |  |  |  |  |  |  | 1.18 |

17. Secondary Outcome: Clearance of Camidanlumab Tesirine
Description: Clearance of HuMax-TAC, PBD-conjugated HuMax-TAC, and free warhead (SG3199).
Time Frame: Pre-dose on Day 1 and 1 to 336 hours post-dose of Cycles 1 and 2 (21 day cycle length)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/day
Arm/Group | 3 μg/kg | 5 μg/kg | 8 μg/kg | 13 μg/kg | 20 μg/kg | 30 μg/kg | 45 μg/kg | 60 μg/kg | 80 μg/kg | 100 μg/kg | 150 μg/kg | 300 μg/kg
Number analyzed (Participants) | 0 | 0 | 2 | 2 | 1 | 18 | 33 | 23 | 18 | 2 | 2 | 1
Liters/day
  Cycle 1 - HuMax-TAC: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 23 | 23 | 18 | 2 | 2 | 1
  Cycle 1 - HuMax-TAC |  |  |  |  |  | 1.82 (69.0) | 1.29 (64.0) | 1.24 (54.5) | 1.60 (184) | 1.82 (136) | 1.05 (22.6) | 0.489
  Cycle 2 - HuMax-TAC: number analyzed (Participants) | 0 | 0 | 2 | 2 | 1 | 18 | 33 | 23 | 15 | 1 | 2 | 1
  Cycle 2 - HuMax-TAC |  |  | 3.23 (50.1) | 1.44 (22.5) | 2.01 | 1.60 (66.5) | 1.03 (61.2) | 0.950 (85.9) | 1.10 (46.2) | 0.446 | 0.849 (30.8) | 1.23
  Cycle 1 - PBD-conjugated HuMax-TAC: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 7 | 29 | 19 | 17 | 2 | 2 | 1
  Cycle 1 - PBD-conjugated HuMax-TAC |  |  |  |  | 0.943 | 1.75 (55.6) | 1.68 (50.3) | 1.65 (48.9) | 1.87 (99.0) | 1.94 (98.7) | 1.33 (18.4) | 0.643
  Cycle 2 - PBD-conjugated HuMax-TAC: number analyzed (Participants) | 0 | 0 | 1 | 2 | 1 | 18 | 33 | 23 | 17 | 2 | 2 | 1
  Cycle 2 - PBD-conjugated HuMax-TAC |  |  | 3.27 | 1.79 (25.1) | 2.46 | 1.93 (57.2) | 1.37 (55.3) | 1.27 (62.8) | 1.44 (86.9) | 3.28 (2602) | 1.17 (15.0) | 1.38
  Cycle 2 - Free warhead (SG3199): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Cycle 2 - Free warhead (SG3199) |  |  |  |  |  |  |  |  |  |  | 4302 |

18. Secondary Outcome: Number of Participants With Anti-drug Antibody Response (ADA) Against Camidanlumab Tesirine
Description: An assay determines the presence of anti-ADCT-301 antibodies in human serum using a validated bridging electro chemiluminescence immunoassay (ECLIA) technique. The technique uses the drug itself to capture any anti ADCT-301 antibodies present in the serum. If anti-ADCT-301 antibodies are detected, they are confirmed to be specifically against ADCT-301 and then the level of the anti-ADCT-301 antibodies present in the serum is established using a modified version of the ECLIA technique.
Time Frame: as for outcome 6
Population: Safety Analysis Set - The safety analysis set consisted of all participants who received camidanlumab tesirine.
Measure: Count of Participants; unit: Participants
Arm/Group | 3 μg/kg | 5 μg/kg | 8 μg/kg | 13 μg/kg | 20 μg/kg | 30 μg/kg | 45 μg/kg | 60 μg/kg | 80 μg/kg | 100 μg/kg | 150 μg/kg | 300 μg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 3 | 2 | 20 | 41 | 29 | 26 | 3 | 2 | 1
Participants
  Confirmed positive ADA pre-dose | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Confirmed positive ADA post-dose only | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Confirmed positive ADA at any time | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to 84 days after last dose (median time on treatment was 43 days [min 1 day; max 354 days])
Description: AEs and SAEs were collected from Day 1 to 84 days after last dose (median time on treatment was 43 days [min 1 day; max 354 days]). All cause mortality was collected from Day 1 to End of Study (maximum of 12 months after last dose; median time on treatment was 43 days [min 1 day; max 354 days]).
Arm/Group | 3 μg/kg | 5 μg/kg | 8 μg/kg | 13 μg/kg | 20 μg/kg | 30 μg/kg | 45 μg/kg | 60 μg/kg | 80 μg/kg | 100 μg/kg | 150 μg/kg | 300 μg/kg
All-Cause Mortality (participants affected / at risk) | 1/2 | 1/2 | 2/2 | 2/3 | 1/2 | 3/20 | 11/41 | 15/29 | 15/26 | 3/3 | 1/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/2 | 0/2 | 3/3 | 1/2 | 10/20 | 24/41 | 14/29 | 18/26 | 1/3 | 1/2 | 1/1
Other Adverse Events (participants affected / at risk) | 1/2 | 2/2 | 2/2 | 3/3 | 2/2 | 20/20 | 41/41 | 29/29 | 26/26 | 3/3 | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 μg/kg (N=2) | 5 μg/kg (N=2) | 8 μg/kg (N=2) | 13 μg/kg (N=3) | 20 μg/kg (N=2) | 30 μg/kg (N=20) | 45 μg/kg (N=41) | 60 μg/kg (N=29) | 80 μg/kg (N=26) | 100 μg/kg (N=3) | 150 μg/kg (N=2) | 300 μg/kg (N=1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spleen disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 6 (7) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hodgkins disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (5) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3 μg/kg (N=2) | 5 μg/kg (N=2) | 8 μg/kg (N=2) | 13 μg/kg (N=3) | 20 μg/kg (N=2) | 30 μg/kg (N=20) | 45 μg/kg (N=41) | 60 μg/kg (N=29) | 80 μg/kg (N=26) | 100 μg/kg (N=3) | 150 μg/kg (N=2) | 300 μg/kg (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1 | 6 | 8 | 2 | 5 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 2 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 8 | 8 | 7 | 7 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 5 | 12 | 3 | 4 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 11 | 3 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 5 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 4 | 4 | 1 | 5 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 5 | 2 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 2 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Lip blister (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 1 | 0 | 10 | 16 | 13 | 7 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 11 | 8 | 8 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 4 | 5 | 4 | 5 | 1 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 2 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 1 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 3 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspergillus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 3 | 8 | 8 | 6 | 1 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 9 | 6 | 4 | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 6 | 6 | 1 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 6 | 5 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 4 | 8 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 3 | 6 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 5 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 2 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 8 | 6 | 2 | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 0 | 2 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 3 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 2 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 7 | 2 | 5 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 1 | 5 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 4 | 2 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 5 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 4 | 2 | 4 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 3 | 2 | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 4 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 5 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 3 | 2 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 5 | 9 | 6 | 7 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 7 | 6 | 4 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 3 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 3 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 7 | 16 | 9 | 4 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 9 | 4 | 4 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 7 | 5 | 5 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 5 | 5 | 2 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 4 | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 2 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can publish after first multi-site publication or if no multi-site publication is made within 18 months of study completion/termination. The only disclosure restriction on PI is sponsor can review results comms. prior to public release and can embargo comms. regarding trial results for a period >60 but ≤180 days from time submitted to sponsor review. Sponsor can't require changes to the comms, extend embargo or require changes to comms, except removing confidential info that are not results

DOCUMENTS (2):
  • Study Protocol (2019-01-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT02432235/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/35/NCT02432235/SAP_001.pdf